CLINICAL TRIAL: NCT00907361
Title: The MagnaSafe Registry: Determining the Risks of MRI in the Presence of Pacemakers and Implantable Cardioverter Defibrillators
Brief Title: The MagnaSafe Registry: Determining the Risks of Magnetic Resonance Imaging (MRI) in the Presence of Pacemakers and Implantable Cardioverter Defibrillators (ICDs)
Acronym: MagnaSafe
Status: Completed | Type: Observational
Sponsor: Scripps Health (Other)
Collaborators: Scripps Clinic (Other); Abbott Medical Devices (Industry); Boston Scientific Corporation (Industry); Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MagnaSafe-095151
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Need for MRI Imaging With Pacemaker or; Implantable Cardioverter Defibrillator Implanted
Keywords: pacemaker; ICD; Implantable Cardioverter Defibrillator; MRI; Magnetic Resonance Imaging
MeSH Terms: interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MRI with pacemaker or ICD — The aim of the present protocol is to prospectively determine the adverse event rate of non-thoracic MRI for patients with implanted cardiac devices by collecting pre- and post-MRI device interrogations in a multi-center registry.

SUMMARY:
This study will create a registry of patients with pacemakers and implantable ICDs who will undergo clinically indicated MRI and will document the incidence of any adverse events or changes in device parameters that might be associated with the procedure.

DETAILED DESCRIPTION:
The MagnaSafe Registry is an investigator initiated study designed to determine the risks of performing MRI for patients with pacemakers and Implantable Cardioverter-Defibrillators (ICDs). We hope that the results of the registry will provide physicians the risk-assessment data needed to assess the use of MRI as a diagnostic tool when no alternative diagnostic imaging technology is appropriate.

The number of patients living with permanent pacemakers or ICD devices in the United States is increasing dramatically as a result of expanded indications. Between 1990 and 2005, an estimated 2.8 million pacemakers and 690,000 ICDs were implanted in the United States. The number of implanted devices continues to increase without an apparent plateau.

Magnetic resonance is the imaging modality of choice for the diagnosis of many diseases of the brain, spinal cord, and musculoskeletal system. For some disease states, no acceptable alternative diagnostic imaging method is available. As the number of implanted cardiac devices is increasing, the clinical indications for MRI are expanding as well. Marketing research estimates that approximately 27.5 million MRI procedures were completed in 2007 (The Medical Information Division of IMV, LTD). It is predicted that there is a 50-75% probability that a patient with a pacemaker or ICD will have the need for an MRI over the lifetime of the device.

Most physicians consider the presence of a pacemaker or ICD to be an absolute contraindication to an MRI study. Patients are denied the examination, even when MR is clearly the superior diagnostic modality or when there is no acceptable alternative imaging test available. To provide optimal care to the increasing number of patients with an implanted cardiac device, health care professionals must have the capability to perform MR imaging with minimal risk and full knowledge of the possible complications.

The present study will create a registry of patients with pacemakers and ICDs who will undergo clinically indicated MRI and will document any adverse event or change in device parameters that may be associated with the imaging procedure. The results of this registry will provide the medical community with an accurate documentation of risk to patients and will establish a protocol of patient screening and device reprogramming for the purpose of maximizing the safe performance of MRI as a diagnostic tool in patients with implantable cardiac devices when indicated.

This is a physician-initiated study that will be coordinated by Scripps Clinic, Green Hospital. It is being performed under an IDE from the FDA. Funding for the MagnaSafe Registry comes from multiple sources including competitive grants, institutional grants, foundation fellowship support, unrestricted educational grants from industry, and philanthropy.

Scripps Clinic/Green Hospital, La Jolla, CA, has performed more than 125 MRIs on patients with implanted cardiac devices. Results of retrospective clinical observations at Scripps Clinic were presented at the American Heart Association 2008 Scientific and American College of Cardiology 2009 Scientific Sessions.

Up to 35 sites will be recruited to participate in the registry. The registry uses a protocol designed to minimize potential risk to the patient and device. MRI compatible equipment will be required to monitor vital signs (non-invasive blood pressure monitoring, pulse oximeter, and single lead cardiac rhythm monitor) while performing scans on patients with implanted devices. Recommendations from the American Heart Association for performance of MR examination in patients with pacemakers or ICDs will be followed.

The MRI procedures will be conducted for clinical purposes at the discretion of the ordering physician. MR examination of patients with permanent implanted cardiac devices will only be performed if there are highly compelling circumstances and when the benefits clearly outweigh the risks in the opinion of the ordering physician. The decision to have an MRI must be based on clinical indication, and is not part of the research protocol.

Those wishing to participate in the registry as an investigational site will be required to obtain approval of the FDA-authorized protocol from their reviewing IRB, and complete a written investigator agreement.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older
* Able to provide informed consent
* Permanent implanted pacemaker or ICD
* Strong clinical indication for MRI; in the clinical setting where MRI is the diagnostic modality of choice for a specific disease state without acceptable alternative imaging technology as determined by the ordering physician.
* Patient is scheduled for non-thoracic MRI (joint, extremity, brain, pelvis, cervical, and lumbar or sacral spine)

Exclusion Criteria:

* Metallic objects that represent a contraindication to MR imaging, including: intra-orbital or intra-ocular retained metal fragments, and intracranial vascular clips and coils
* Claustrophobia unresponsive to pre-procedure sedatives
* Morbid obesity (abdominal diameter >60 cm)
* ICD or pacemaker generator placement prior to 2002
* ICD and pacing dependent
* Pregnancy
* Device generator battery voltage at elective replacement index (ERI)
* Presence of active implantable medical device (other than pacemaker or ICD)
* Presence of abandoned leads (with the exception of post CABG temporary epicardial pacing wires)
* Presence of implanted cardiac device in the abdominal position
* Pacemaker or ICD that is labeled as MRI-Conditional (approved by the FDA for exposure to MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with pacemaker or ICD that is scheduled for a clinically indicated MRI.
Sampling Method: Non-Probability Sample
Enrollment: 2039 (Actual)
Dates: Start 2009-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Rate of device failure. | Anytime during follow up

SECONDARY OUTCOMES:
Rate of device parameter changes | Anytime during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Russo, MD, PhD, Principal Investigator — Scripps Clinic
Locations (21):
- United States (21):
  - Providence St. Joseph Medical Center, Burbank, California
  - Scripps Clinic/Green Hospital, La Jolla, California
  - Scripps Memorial Hospital, La Jolla, California
  - UCLA Cardiac Arrhythmia Center, Los Angeles, California
  - Spectrum Clinical Research, Moreno Valley, California
  - University of California, San Diego, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Aventura Hospital and Medical Center, Aventura, Florida
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Providence Heart Institute, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Valley Hospital, Ridgewood, New Jersey
  - Advanced Cardiovascular Imaging, New York, New York
  - Oklahoma Heart Research and Education Foundation, Tulsa, Oklahoma
  - Abington Health System, Abington, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Russo RJ, Costa HS, Silva PD, Anderson JL, Arshad A, Biederman RW, Boyle NG, Frabizzio JV, Birgersdotter-Green U, Higgins SL, Lampert R, Machado CE, Martin ET, Rivard AL, Rubenstein JC, Schaerf RH, Schwartz JD, Shah DJ, Tomassoni GF, Tominaga GT, Tonkin AE, Uretsky S, Wolff SD. Assessing the Risks Associated with MRI in Patients with a Pacemaker or Defibrillator. N Engl J Med. 2017 Feb 23;376(8):755-764. doi: 10.1056/NEJMoa1603265. PMID 28225684
- [Derived] Wiesenfeld HC. Screening for Chlamydia trachomatis Infections in Women. N Engl J Med. 2017 Feb 23;376(8):765-773. doi: 10.1056/NEJMcp1412935. No abstract available. PMID 28225683